CLINICAL TRIAL: NCT05170425
Title: Observational Registry Study With Sub-analysis (Patients Previously Randomized to LAMBDA 001) to Assess ProsperaTM Performance for Detection of CLAD After Lung Transplant (LAMBDA 002)
Brief Title: LAMBDA 002 (Lung Registry) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-055-TRP
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lung Transplant Rejection
Keywords: Prospera; Lung Transplant; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: 1) Cohort 1: Previously enrolled AND randomized in LAMBDA 001 Participants enrolled to Cohort 1 will be enrolled at least 12 and up to 18 months post-transplant.
  Interventions: Device: Prospera
- Cohort 2: 2) Cohort 2: Not previously randomized in LAMBDA 001 Participants who were enrolled in LAMBDA 001 but who were not randomized in LAMBDA 001 may be enrolled to Cohort 2.
  Interventions: Device: Prospera

INTERVENTIONS:
Device: Prospera — Prospera™ detects allograft rejection noninvasively and with high accuracy by measuring the fraction of donor derived cell-free DNA (dd-cfDNA) in the patient's blood, without the need for prior donor or recipient genotyping.
  Prospera is a commercially available Laboratory Developed Test (LDT) certified under the Clinical Laboratory Improvement Amendments (CLIA). This test has not been cleared or approved by the U.S. Food and Drug Administration (FDA).

SUMMARY:
The LAMBDA 002 registry study is an observational, longitudinal, multi-center study observing patients undergoing lung transplant.

DETAILED DESCRIPTION:
The LAMBDA 002 registry study is an observational, longitudinal, multicenter study observing patients undergoing lung transplant in one of the following two cohorts:

Cohort 1: Previously enrolled and randomized in LAMBDA 001 (transbronchial biopsy surveillance or Prospera surveillance) and enrolled at least 12 and up to 18 months post-transplant.

Cohort 2: Not previously randomized in LAMBDA 001 (may have been enrolled but randomization did not occur), Prospera testing is part of clinical care and enrolled during less than or equal to 12 months posttransplant.

Primary Objective:

The primary objective of the study is to assess the clinical utility of combining Prospera testing with routine transplant management in detecting acute rejection or infection events in patients receiving Prospera testing as part of their post-transplant clinical care.

Secondary Objectives:

The secondary objectives of the study are to:

1. Determine whether Prospera can detect AR (acute rejection) and/or infection earlier than standard clinical indicators used concurrently during the study.
2. Evaluate Prospera's ability to differentiate between rejection and infectious injuries for single and repeat episodes of bacterial, viral, mycobacterial and fungal infections.
3. Evaluate changes in Prospera dd-cfDNA as an indicator for biopsy proven acute rejection (BPAR), graft failure, death, development of donor-specific antibodies (DSA), chronic lung allograft dysfunction (CLAD), infection episodes and response to treatment for rejection.
4. Evaluate changes in Prospera dd-cfDNA in assessments involving standard management for acute rejection and infection events.

ELIGIBILITY:
Patients must meet all the following selection criteria to be eligible for the study:

Inclusion Criteria

1. Age 18 or older at the time of enrollment.
2. Underwent a first single or bilateral deceased-donor lung transplant. 3) Allograft was from a genetically different donor (e.g., not an identical twin).

4) Meets criteria for one of the two study cohorts:

a) Cohort 1: i) Previously enrolled and randomized in LAMBDA 001 (TBBx surveillance or Prospera surveillance) AND ii) Enrolled at least 12 and up to 18 months post-transplant b) Cohort 2: i) Not previously randomized in LAMBDA 001 (may have been enrolled if randomization did not occur) AND ii) Enrolled less than or equal to 12 months post-transplant 5) Prospera testing is planned as part of routine post-transplant management.

Exclusion Criteria

Patients are not eligible for the study if they meet any of the following criteria:

1) Recipient of multi-organ transplant at the time of lung transplant. 2) Prior recipient of any solid organ or hematopoietic (bone marrow or stem cell) transplant.

3) Human immunodeficiency virus (HIV) infection. 4) Pregnant. 5) Ongoing testing with another allograft dd-cfDNA assessment test is planned. 6) Unwilling or unable to provide informed consent. 7) Unwilling or unable to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung Transplantation Patient
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percent of donor-derived cell-free DNA (ddcfDNA) measured via the Prospera test | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Ross, MD, Principal Investigator — Natera, Inc.
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, California City, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Corewell Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Washington, Seattle, Washington